CLINICAL TRIAL: NCT06551753
Title: Distraction-Based Interventions During Implanted Venous Port Catheter Needle Entry: Virtual Reality Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Esra ibek, Oncology Clinic Nurse, Uludag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UÜEİ001
Record Dates: First submitted 2024-07-14; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: a randomized controlled experimental study
Masking Description: Given the nature of the intervention, the investigator and patients were not blinded to the intervention. Since the patients in the intervention group were fitted with virtual reality glasses, blinding could not be performed due to the nature of the study. However, patients were blind to randomization until administration began. After the patient was pre-tested, he was informed by the researcher that he was in the intervention or control group. The investigator was also blind to randomization. Patients were assigned to intervention and control groups by an independent selection from a simple bag of random numbers prepared for randomization. Analysis of the study data was also performed by an independent statistician who was unaware of the intervention and control groups. In this study, blinding was ensured in the implementation of randomization and analysis and reporting of data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- virtual reality app (Experimental): virtual reality app
  Interventions: Other: virtual reality app

INTERVENTIONS:
Other: virtual reality app — virtual reality app

SUMMARY:
This study is a randomized controlled experimental study planned to examine the effect of virtual reality application during implanted venous port catheter needle insertion on patient satisfaction, comfort level and time perception in cancer patients. Distraction-based interventions used in symptom management of cancer patients are simple, effective and cost-effective. Distraction applications such as virtual reality glasses, listening to music, painting and daydreaming aim to focus attention on another stimulus. Virtual reality application uses human-machine interfaces to focus the patient on a world other than their current environment with a three-dimensional virtual video, changing their perception of space and time. It has been shown that virtual reality applications reduce pain and anxiety, increase patient satisfaction, provide relief, and positively affect vital parameters during procedural procedures such as bone marrow aspiration, fine needle aspiration breast biopsy, colonoscopy, and transrectal prostate biopsy in cancer patients receiving chemotherapy.

Virtual reality is a new technique developed thanks to the advancement of computer technology and started to be used in the field of health as a cognitive-behavioral method to relieve pain and relax the patient. This method uses human-machine interfaces to give people the feeling of being in an interactive environment with virtual video in the forest, ocean or space. Virtual reality glasses are an application that is used to isolate the patient from his/her environment and includes a distraction method that allows the patient to focus on another world in three dimensions. It is usually applied with glasses or headgear. In addition, the patient is prevented from perceiving the surrounding sounds by wearing headphones. The most important feature that distinguishes virtual reality from other technological products such as television and video games is that it gives users the feeling of being in a different place. The use of virtual reality glasses provides a positive environment for patients and provides a calming experience by changing their perception of time.Virtual reality applications, a new technology, can make a positive difference in cancer care and increase the comfort and satisfaction levels of cancer patients. This innovative method can be used as a complementary nursing approach in addition to standard care during implantable venous port catheter needle intervention. The widespread use of virtual reality applications in cancer care contributes to qualified nursing care. This study will be presented as an innovative method showing that virtual reality technologies can be incorporated into nursing practices.

DETAILED DESCRIPTION:
This study is a randomized controlled experimental study planned to examine the effect of virtual reality application during implanted venous port catheter needle insertion on patient satisfaction, comfort level and time perception in cancer patients. Distraction-based interventions used in symptom management of cancer patients are simple, effective and cost-effective. Distraction applications such as virtual reality glasses, listening to music, painting and daydreaming aim to focus attention on another stimulus. Virtual reality application uses human-machine interfaces to focus the patient on a world other than their current environment with a three-dimensional virtual video, changing their perception of space and time. It has been shown that virtual reality applications reduce pain and anxiety, increase patient satisfaction, provide relief, and positively affect vital parameters during procedural procedures such as bone marrow aspiration, fine needle aspiration breast biopsy, colonoscopy, and transrectal prostate biopsy in cancer patients receiving chemotherapy.

Virtual reality is a new technique developed thanks to the advancement of computer technology and started to be used in the field of health as a cognitive-behavioral method to relieve pain and relax the patient. This method uses human-machine interfaces to give people the feeling of being in an interactive environment with virtual video in the forest, ocean or space. Virtual reality glasses are an application that is used to isolate the patient from his/her environment and includes a distraction method that allows the patient to focus on another world in three dimensions. It is usually applied with glasses or headgear. In addition, the patient is prevented from perceiving the surrounding sounds by wearing headphones. The most important feature that distinguishes virtual reality from other technological products such as television and video games is that it gives users the feeling of being in a different place. The use of virtual reality glasses provides a positive environment for patients and provides a calming experience by changing their perception of time. Virtual reality applications, a new technology, can make a positive difference in cancer care and increase the comfort and satisfaction levels of cancer patients. This innovative method can be used as a complementary nursing approach in addition to standard care during implantable venous port catheter needle intervention. The widespread use of virtual reality applications in cancer care contributes to qualified nursing care. This study will be presented as an innovative method showing that virtual reality technologies can be incorporated into nursing practices.

Research Inclusion Criteria:

* Those between the ages of 18-65
* Those receiving active chemotherapy
* Those who volunteer to participate in the research
* Having an implantable venous port catheter
* Those who will use virtual reality glasses for the first time

Exclusion Criteria from the Research:

* Presence of metastasis
* Those receiving anxiolytic drug treatment
* Those receiving antidepressant medication
* People with communication, hearing and vision problems
* Having any psychiatric disorder
* Those who used any analgesic medication at least 8 hours before
* Those with migraine, vertigo, active nausea-vomiting, headache, dizziness problems Patient introductory information form, satisfaction status evaluation scale, general comfort scale-short form and time perception evaluation form during the procedure will be used as data collection tools.

Data Collection Phase:

Before starting the research, written informed consent will be obtained from cancer patients who agree to participate in the study and meet the inclusion criteria, by explaining the purpose and rationale of the research. In the research, simple randomization method will be used to determine the sample number of intervention and control groups. They will be assigned to the control (n = 35) and intervention (n = 35) groups by simple randomization method from a simple random numbers table prepared before the study. Using the simple random numbers table, patients assigned to the intervention group will be shown a three-minute video, determined by the patient's choice, from video scenes containing nature images with sound shot at a 360-degree angle recorded on YouTube, through a virtual reality headset, throughout the procedure. The application will begin as soon as the patient is positioned, just before the procedure begins, and will continue after the procedure is completed, allowing them to experience a three-dimensional virtual reality application that lasts approximately 3 minutes. Data will be collected by face-to-face interview with patients before and after the procedure. Patient introductory information form, satisfaction status evaluation scale, general comfort scale-short form and time perception evaluation form during the procedure will be used as data collection tools. The study will be carried out in the same environment with a single nurse, the same measurement tools will be used, and procedures will be applied to both the control and experimental groups by the same nurse.

Evaluation of Data:

Descriptive and comparative statistics, correlation and regression analyzes will be used to evaluate the data obtained from the study. SPSS 25.0 Package Program will be used to analyze the data. Categorical measurements will be presented as numbers and percentages, and numerical measurements will be presented as mean and standard deviation, median, minimum and maximum values. Chi-Square Test statistics will be used to compare categorical measurements between groups. Whether numerical measurements provide normal distribution will be evaluated with the Kolmogrov-Smirnov Test. In independent groups, t test will be used, and if the assumptions are not met, Mann Whitney U test will be used. Spearman correlation analyzes will be applied for correlation analyzes between data. Statistical significance level will be accepted as p<0.05. The research results will be evaluated and presented in the light of the literature.

CENTER/CENTERS WHERE THE RESEARCH WILL BE CONDUCTED; Bursa Uludağ University Faculty of Medicine Hospital Medical Oncology Polyclinic

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18-65
* Those receiving active chemotherapy
* Those who volunteer to participate in the research
* Having an implantable venous port catheter
* Those who will use virtual reality glasses for the first time

Exclusion Criteria:

* Presence of metastasis
* Those receiving anxiolytic drug treatment
* Those receiving antidepressant medication
* People with communication, hearing and vision problems
* Having any psychiatric disorder
* Those who used any analgesic medication at least 8 hours before
* Those with migraine, vertigo, active nausea-vomiting, headache, dizziness problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-07-13 (Actual)

PRIMARY OUTCOMES:
beginning | Before port needle placement
  Before the procedure, patient information form, satisfaction assessment scale, general comfort scale-short form were filled out in both groups.

SECONDARY OUTCOMES:
finish | after port needle placement
  After the procedure was completed, the satisfaction evaluation scale, general comfort scale-short form and time perception evaluation form during the procedure were filled out.

CONTACTS AND LOCATIONS:
Overall Officials: Derya Çınar, Doç. Dr., Study Director — Izmir Bakircay University
Locations (1):
- İzmir Bakırçay University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen YB, Bao HS, Hu TT, He Z, Wen B, Liu FT, Su FX, Deng HR, Wu JN. Comparison of comfort and complications of Implantable Venous Access Port (IVAP) with ultrasound guided Internal Jugular Vein (IJV) and Axillary Vein/Subclavian Vein (AxV/SCV) puncture in breast cancer patients: a randomized controlled study. BMC Cancer. 2022 Mar 5;22(1):248. doi: 10.1186/s12885-022-09228-6. PMID 35248019
- [Background] Brunetti GA, Tendas A, Meloni E, Mancini D, Maggiore P, Scaramucci L, Giovannini M, Niscola P, Cartoni C, Alimena G. Pain and anxiety associated with bone marrow aspiration and biopsy: a prospective study on 152 Italian patients with hematological malignancies. Ann Hematol. 2011 Oct;90(10):1233-5. doi: 10.1007/s00277-011-1166-7. Epub 2011 Feb 2. No abstract available. PMID 21287348
- [Background] Taxbro K, Hammarskjold F, Thelin B, Lewin F, Hagman H, Hanberger H, Berg S. Clinical impact of peripherally inserted central catheters vs implanted port catheters in patients with cancer: an open-label, randomised, two-centre trial. Br J Anaesth. 2019 Jun;122(6):734-741. doi: 10.1016/j.bja.2019.01.038. Epub 2019 Apr 17. PMID 31005243
- [Background] Schirrmacher V. From chemotherapy to biological therapy: A review of novel concepts to reduce the side effects of systemic cancer treatment (Review). Int J Oncol. 2019 Feb;54(2):407-419. doi: 10.3892/ijo.2018.4661. Epub 2018 Dec 10. PMID 30570109
- [Background] Gupta A, Scott K, Dukewich M. Innovative Technology Using Virtual Reality in the Treatment of Pain: Does It Reduce Pain via Distraction, or Is There More to It? Pain Med. 2018 Jan 1;19(1):151-159. doi: 10.1093/pm/pnx109. PMID 29025113
- [Background] Hundert AS, Birnie KA, Abla O, Positano K, Cassiani C, Lloyd S, Tiessen PH, Lalloo C, Jibb LA, Stinson J. A Pilot Randomized Controlled Trial of Virtual Reality Distraction to Reduce Procedural Pain During Subcutaneous Port Access in Children and Adolescents With Cancer. Clin J Pain. 2021 Dec 30;38(3):189-196. doi: 10.1097/AJP.0000000000001017. PMID 34974512